CLINICAL TRIAL: NCT00298909
Title: Exercise Versus Extended-Release Niacin in Patients With Coronary Heart Disease and Low High-Density Lipoproteins (HDL) Cholesterol: Effect on Lipid Profile and Endothelial Function
Brief Title: Exercise Versus Niacin in Patients With Coronary Artery Disease (CAD) and Low High-Density Lipoproteins (HDL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Steffen Desch, MD, Priv.-Doz. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Leipzig-02
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Disease; Hypolipoproteinemia
MeSH Terms: conditions — Coronary Disease; Hypolipoproteinemias | interventions — Exercise; Niacin

ARMS (3):
- 1 (Experimental): niacin
  Interventions: Drug: niaspan (extended-release niacin); Drug: niacin
- 2 (Active Comparator): physical exercise
  Interventions: Behavioral: physical exercise
- 3 (Placebo Comparator): control
  Interventions: Other: control

INTERVENTIONS:
Behavioral: physical exercise — physical exercise
  Arms: 2
Drug: niaspan (extended-release niacin) — niaspan (extended-release niacin)
  Arms: 1
Drug: niacin — niacin extended-release
  Arms: 1
Other: control — control
  Arms: 3

SUMMARY:
The investigators want to study the relative effects of physical exercise vs. extended-release niacin (lipid-lowering drug) in patients with coronary heart disease and low HDL cholesterol ("good cholesterol") on

* lipid profile
* endothelial function as measured by ultrasound

The endothelium is the inner part of the blood vessels. Impaired endothelial function is known to be associated with atherosclerosis which can ultimately lead to diseases such as stroke, heart attack and others. Endothelial function can be assessed non-invasively by ultrasound.

Both interventions mentioned above have been shown to have a beneficial effect on lipid profile and endothelial function. However, the relative effects are unclear.

DETAILED DESCRIPTION:
Comparison of physical exercise vs. extended-release niacin in patients with CAD and low HDL cholesterol (< 1,03 mmol/L) on lipid profile and endothelial function as measured by flow-mediated dilatation of radial artery. Secondary goals are the assessment of biochemical markers of atherosclerosis, expression of monocyte surface markers, oxidative stress and thrombogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Coronary disease
* Low HDL cholesterol
* Age limits (see below)

Exclusion Criteria:

* Unstable angina oder MI within 3 months prior to inclusion
* CAD with indication for bypass surgery
* Left main disease ( > 25% stenosis diameter)
* Ejection fraction < 40%
* Higher degree heart valve disease
* Higher degree ventricular arrhythmias
* Type 1 Diabetes
* Severe disorders of lipoprotein metabolism (Low-density lipoprotein cholesterol (LDL)> 5.0 mmol/L)
* Severe liver disease
* Thyroid disease
* Alcohol or drug abuse
* Pregnancy
* Stroke or Transient Ischemic Attack (TIA) within 3 months prior to inclusion
* Allergy against niacin oder other ingredient of niaspan
* Participation in other clinical trial within 30 days prior to inclusion
* Acute gastric ulcer
* Arterial bleeding
* Uncontrolled severe arterial hypertension
* Treatment with lipid-lowering drug other than Hydroxy-Methylglutaryl Coenzyme A (HMG-CoA)-inhibitor within 3 months prior to inclusion

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
relative effect on flow-mediated dilatation of radial artery | 6 months

SECONDARY OUTCOMES:
lipid profile | 6 months
biochemical markers of atherosclerosis | 6 months
expression of monocyte surface markers | 6 months
oxidative stress | 6 months
thrombogenicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Desch, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig Heart Center, Leipzig, Germany